CLINICAL TRIAL: NCT04411329
Title: Caudal Epidural With Non Opioid Adjuvants in Lumbosacral Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sanaa Farag Mahmoud Wasfy, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R15/2020
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Caudal Analgesia for Lumosacral Spine Surgeries
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): patients will receive 30 ml of 0.125% bupivacaine with 8 mg dexamethasone (20 ml before skin incision and 10 ml at end of surgery
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone
- group B (Active Comparator): we will add 50µg dexmedetomidine to the previous mixture given to group A (20 ml before skin incision and 10 ml at end of surgery
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone; Drug: Dexmedetomidine
- group c (Active Comparator): we will add 1500 IU hyalurodinase to the mixture given to group A. (20 ml before skin incision and 10 ml at end of surgery
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone; Drug: Hyalouridinase

INTERVENTIONS:
Drug: Bupivacaine — local anesthetics, steriod, alpha 2 blockers
Drug: Dexamethasone — dexamethazone
Drug: Dexmedetomidine — dexmedetomidine
  Arms: group B
Drug: Hyalouridinase — hyalouridinase
  Arms: group c

SUMMARY:
Lumbosacral spine surgeries are accompanied with severe postoperative pain which has a negative effect on patients' recovery. Preemptive analgesia before lumbosacral spine surgeries should be implemented to prevent CNS plasticity and to provide effective pain relief.

The most common way to provide pain management after spine surgery is the intravenous analgesia. Caudal epidural analgesia can be a highly effective method for postoperative pain relief.

The most common way to provide pain management after spine surgery is the intravenous analgesia. Caudal epidural analgesia can be a highly effective method for postoperative pain relief. acting drugs last from 4-8 hours,But this can be prolonged by adding non opioid adjuvants like steroid( dexamethazone,betamethasone), alpha2 agonists (clonidine, dexmedetomidine), or their combination. This study will compare adding different non opioid adjuvants to bupivacaine in caudal epidural for preventive analgesia in lumbosacral spine surgery which can be a part of multimodal analgesia protocol.

.

DETAILED DESCRIPTION:
60 patient will be enrolled in the study. They will be allocated randomly into 3 groups. after induction of general anesthesia and changing the patient into prone position injection of the study cocktail through caudal epidural route.(20 ml before skin incision and 10 ml of the same mixture at the end of surgery) in all patients.

In the first group patients will receive 0.125% bupivacaine with 8 mg dexamethasone In the second group we will add 50µg dexmedetomidine to the previous mixture given to the first group.

In the third group we will add 1500 IU hyalurodinase to the mixture given to the first group

During the operation adjustment of sevoflurane concentration and fentanyl incremental doses (0.5 μg/kg) will be according to hemodynamic measurements.

Clinical signs of inadequate analgesia is defined as an increase in blood pressure and heart rate more than 20% from baseline. Efficacy of the caudal epidural block will be tested at beginning of skin incision (15-20 minutes after block). If signs of inadequate analgesia are observed, fentanyl 0.5 µg/kg will be given and those patients will be excluded from the study.

In case of decrease in Blood Pressure greater than 20% from baseline, the patient will be infused by 500 ml ringer lactate and if blood pressure is not responding, administration of increments of 3 mg ephedrine will be given. Also If heart rate decreased to 45 beats/min, atropine sulfate 0.01 mg/kg will be given. Muscle paralysis will be antagonized by sugmmadex 2mg/kg at the end of surgery after switching the patient to the supine position.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged from 18-65 years , ASA I and II, scheduled for lumbar spine surgery (laminectomy, discectomy, foraminotomy, fenestration or fusion) in a virgin back.

Exclusion Criteria:

* Patients with multiple level fixation, revision surgery, complicated spinal canal stenosis, traumatic lumbar surgeries were excluded, patients with addiction, allergy to local anesthetics or to any drug used in the study and those with coagulation abnormality are also excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia | postoerative 24 hours.
  time from second dose caudal epidural block to first analgesic requirement

SECONDARY OUTCOMES:
postoperative pain | postoperative 24 hours
  VAS score from zero for (no pain) till 10 for ( the most severe intractable pain)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sanaa Farag Mahmoud, Cairo, New Cairo
  - Ainshams hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solanki SL, Bharti N, Batra YK, Jain A, Kumar P, Nikhar SA. The analgesic effect of intrathecal dexmedetomidine or clonidine, with bupivacaine, in trauma patients undergoing lower limb surgery: a randomised, double-blind study. Anaesth Intensive Care. 2013 Jan;41(1):51-6. doi: 10.1177/0310057X1304100110. PMID 23362890
- [Background] Barham G, Hilton A. Caudal epidurals: the accuracy of blind needle placement and the value of a confirmatory epidurogram. Eur Spine J. 2010 Sep;19(9):1479-83. doi: 10.1007/s00586-010-1469-8. Epub 2010 May 29. PMID 20512512